CLINICAL TRIAL: NCT05424263
Title: The Short-chain Fatty Acid Acetate for Improving Age-associated Arterial Dysfunction
Brief Title: Acetate and Age-associated Arterial Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0473
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Aging; Vascular Stiffness; Vascular Dilation
Keywords: Acetate; Short-chain fatty acids; Gut microbiome; Arterial function
MeSH Terms: interventions — calcium acetate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. The study drug and placebo will be compounded into visually-identical oral liquid solutions and packaged in identical opaque brown medicine bottles. Only the pharmacy and biostatistician conducting the randomization will know which group subjects are assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetate (Experimental): Subjects will be orally supplemented with calcium acetate for 12 weeks. Subjects will be instructed to take a volume of the oral liquid solution that contains 1,334 mg of calcium acetate 3x per day with meals, for a total dose of 4,000 mg/day. Calcium acetate will be compounded by the CU Anschutz Medical Campus Research Pharmacy and dispensed to subjects in 4-week supplies.
  Interventions: Drug: Calcium Acetate Oral Solution
- Placebo (Placebo Comparator): Subjects will be orally supplemented with calcium carbonate for 12 weeks. This placebo has been selected to match any potential effects of calcium and phosphate binding of the calcium acetate, i.e., we will isolate the effects of acetate. Subjects will be instructed to take a volume of the oral liquid solution equal to that of the calcium acetate group 3x per day with meals. To match the amount of elemental calcium between calcium acetate and calcium carbonate, this dose of calcium carbonate will contain 833 mg of calcium carbonate, for a total dose of 2,500 mg/day. Calcium carbonate will be compounded by the CU Anschutz Medical Campus Research Pharmacy, visually identical to calcium acetate including the packaging, and dispensed to subjects in 4-week supplies.
  Interventions: Drug: Calcium Carbonate Oral Suspension

INTERVENTIONS:
Drug: Calcium Acetate Oral Solution — Subjects will be supplemented with calcium acetate (4,000 mg/day), as described in the arm/group descriptions, for 12 weeks.
  Other Names: Calcium acetate
  Arms: Acetate
Drug: Calcium Carbonate Oral Suspension — Subjects will be supplemented with calcium carbonate (2,500 mg/day), as described in the arm/group descriptions, for 12 weeks.
  Other Names: Calcium carbonate
  Arms: Placebo

SUMMARY:
Cardiovascular diseases are the leading cause of morbidity and mortality and contribute most to healthcare costs in the U.S. Age is the strongest cardiovascular disease risk factor, with >90% of all deaths from cardiovascular disease occurring in adults >50 years old. The age-associated increased risk of cardiovascular disease is due, in large part, to the development of arterial dysfunction, including endothelial dysfunction and stiffening of the large elastic arteries. Therefore, novel, effective interventions that improve arterial function will have a large public health impact by decreasing the risk of cardiovascular diseases.

The short-chain fatty acid acetate is endogenously produced by the gut microbiome from fermentation of dietary soluble fiber. High-fiber diets reduce risk of cardiovascular diseases, but unfortunately, a low percentage of Americans meet guidelines for adequate dietary fiber intake and, despite nationwide efforts to improve this, trends in fiber intake have not improved over the last 20+ years. Thus, directly supplementing acetate may be a more practical and feasible intervention for effectively improving arterial function in older adults and reducing the risk of cardiovascular diseases.

The investigators will conduct a study to determine the efficacy of 12 weeks of oral supplementation with acetate for improving arterial function in late middle-aged and older (50+ years) adults. They will also assess the safety and tolerability of acetate supplementation in these adults and perform innovative mechanistic analyses to determine how acetate supplementation improves arterial function. The investigators hypothesize that oral acetate supplementation will improve arterial function by decreasing oxidative stress and increasing nitric oxide bioavailability, and also hypothesize that acetate supplementation will be safe and promote high rates of adherence.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel design clinical trial to assess the efficacy of 12 weeks of oral acetate supplementation for improving arterial function in late middle-aged and older (MA/O) adults (50+ years). The primary outcome is brachial artery flow-mediated dilation (FMDba), the gold-standard measure of endothelial function in humans (hypothesis: FMDba will be improved by acetate). The secondary outcome is carotid-femoral pulse wave velocity (CFPWV), the gold-standard measure of large elastic artery stiffness in humans (hypothesis: CFPWV will be reduced by acetate). Various other outcomes will also be measured. All measures will be assessed before and after 12-weeks of supplementation with 4,000 mg/day calcium acetate or placebo.

* Subject Enrollment and Screening: Potential participants will be made aware of the proposed study through various recruitment efforts. Interested participants will contact the research coordinator via phone or email and will be administered a screening form online through the Research Electronic Data Capture (REDCap) system to determine eligibility. REDCap is a secure web-based application designed to support data capture for research studies.
* After hearing a study description and having questions answered by the research coordinator, those eligible and interested in participating in the study will provide written and verbal informed consent, and undergo in-person screening. The investigators plan to consent and screen 88 interested individuals in order to meet the enrollment target of 66 participants (account for an approximately 20% rate of exclusion based on inclusion/exclusion criteria that can only be determined in-person).
* In-person screening will include: review of medical history; physical exam; resting heart rate; resting blood pressure; and a blood draw for metabolic profile, lipid profile, complete blood count, thyroid stimulating hormone, and serum phosphorus. All screening will take place at the Division of Renal Diseases & Hypertension's Clinical Vascular Physiology Core Laboratory, located within the CU Medicine building on the CU Anschutz Medical Campus.
* Participant Randomization: After completing screening, eligible subjects will be randomized to receive either: 1) calcium acetate; or 2) placebo (calcium carbonate), with equal numbers in each group, using a block randomization scheme to balance age group (middle-aged, 50-64 years vs. older, >=65 years) and sex (male vs. female). This trial will be double-blind. Subjects and members of the investigative team involved in the acquisition and analysis of outcomes will be blinded to group assignment.
* Assessment of Study Outcomes: All subjects will undergo testing for all primary, secondary and other outcome measures, as well as assessment of subject characteristics known to effect arterial function, before and after 12-weeks of acetate or placebo supplementation. All measurements will be made after a 12 hour fast from food and caffeine (water allowed) and 24 hours after the last dose of acetate or placebo. All testing will take place in a temperature-controlled laboratory.

Visit 2:

* The Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire will be completed;
* Sleep questionnaire;
* Body composition assessed by Bod Pod and anthropometry.
* Following visit 3, subjects will take home a kit for collecting urine for 24 hours, 3 swabs to collect fecal samples for gut microbiome composition on 3 separate days, a 3-day diet record to monitor nutrient intake, a Actigraph watch to measure physical activity (wear for 3 days), an ambulatory blood pressure monitor (wear for 24-hours; automatic measurements every 20 minutes). Subjects will be provided with written and verbal instructions for proper operation and completion of all these measures. The diet log and monitors will be returned at the next testing visit.

Visit 4:

* Casual blood pressure;
* IV placement and blood sampling;
* Venous endothelial cell collection;
* Measurements of arterial stiffness (carotid-femoral pulse wave velocity, carotid artery compliance);
* Brachial artery FMD with saline (vascular endothelial function);
* Brachial artery FMD after vitamin C infusion (for oxidative stress-mediated suppression of vascular endothelial function).
* Brachial artery dilation to sublingual nitroglycerin (endothelium-independent dilation).
* After completing baseline testing, subjects will begin their assigned intervention (acetate or placebo). Acetate and placebo will be compounded by the CU Anschutz Pharmacy into identical oral liquid solutions, packaged into opaque brown medicine bottles, and dispensed to subjects in 4-week supplies. The subject's name and instructions for dosing and timing will be labeled on the bottles.

Visits 4-5: Check-in visits (after 2, 4, and 8 weeks on intervention)

* Subjects will discuss any issues with tolerability or treatment-emergent adverse events with the research coordinator **The dose of study drug may be reduced slightly, or the timing of when the drug is taken may be adjusted, if subjects report side effects
* Weigh medicine bottle to determine adherence
* Blood draw for serum phosphate levels, standard clinical blood chemistries, and serum acetate **May repeat 1 week later, after adjusting dose, if any results are abnormal
* On weeks 4 and 8, receive next 4-week supply of study drug

After weeks 1, 6, and 10, the coordinator will check-in with subjects about any issues and treatment-emergent adverse events via phone call.

Post-Testing (Visits 7 & 8):

- After completing 12-weeks of acetate or placebo supplementation, subjects will return to the laboratory for reassessment of all outcome and subject characteristic measures made during visits 2 & 3. Post-testing will be identical to the baseline testing procedures and conditions.

Intervention Duration and Study Sample Size: The expected duration for a participant to complete the entire protocol from screening to follow-up testing is 14-16 weeks. Based on our power analysis, 26 participants per group (acetate vs. placebo; 52 total) are needed to detect a significant difference in our primary outcome measure (FMDba). The investigators intend to enroll 66 subjects (33 per group) to allow for an ~20% dropout rate. Based on this, ~2-3 participants will be enrolled each month.

Data Collection and Analysis (including blinding): Collection of outcome measures data will be performed by the PI, Dr. Vienna Brunt, with the assistance of Amy Bazzoni (research coordinator), other professional research staff at the Clinical Vascular Physiology Core Laboratory and/or trainees within Dr. Brunt's lab. IV placement, blood draws and vascular endothelial cell collection will be performed by an experienced research nurse or nurse practitioner. Processing of endothelial cells and serum exposure experiments will be performed by professional research staff, under the direct supervision of the PI. Data analysis will be performed by Dr. Brunt and/or supervised professional/laboratory research staff. Having a single investigator perform all data collection and analysis will remove the potential for inter-investigator variation. Dr. Brunt will remain blinded throughout data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent;
* Age 50+ years;
* Serum phosphorus levels >= 2.5 mg/dl at screening;
* Habitual dietary fiber intake <30 g/day for men or <21 g/day for women, based on Block Fiber Screener conducted at screening;
* Weight-stable in the 3 months prior to enrollment (self-report);
* Willing to abstain from dietary supplements for 48 hours and from alcohol, tobacco, and cannabis products for 24 hours before all visits;

Exclusion Criteria:

* History of current serious, chronic clinical disease, e.g., cardiovascular disease, diabetes, liver disease, Alzheimer's disease and related dementias, cancer;
* Major changes in health in the past 3 months, e.g., hospitalizations, major surgeries, significant changes in medications;
* Currently taking calcium acetate or any other calcium supplementation;
* Screening FMDba > 8%;
* Body mass index > 40 kg/m^2 at screening;
* Regular vigorous/aerobic endurance >4 bouts/week for >30 min/bout at a workload of >6 METS;
* Any apparent dependence on or abuse of alcohol, tobacco, and cannabis products;
* Pregnancy, breast-feeding, or plans to become pregnant during the duration of the study;
* Any finding on the medical history, physical exam, or standard clinical blood labs that, in the opinion of the physician of record, would put the subject at increased risk with calcium supplementation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Brachial Artery Flow-Mediated Dilation | 12 weeks
  Nitric oxide-mediated endothelium dependent dilation (vascular endothelial function) will be assessed at baseline and end-intervention by flow-mediated dilation of the brachial artery determined using high-resolution ultrasonography (Canon Xario 200) and analyzed with a commercially available software package (Vascular Analysis Tools, Medical Imaging Applications, LLC). Brachial artery flow-mediated dilation will be assessed by measuring brachial artery diameter and forearm blood flow at baseline and for 2 minutes following reactive hyperemia induced by 5 minutes of forearm blood flow occlusion (upper forearm cuff placement). Data will be expressed as a percent change in arterial diameter from pre-cuff inflation diameter, and then as a change in this % from baseline to end-intervention.

SECONDARY OUTCOMES:
Change in Carotid-Femoral Pulse Wave Velocity (CFPWV) | 12 weeks
  A transcutaneous tonometer (Noninvasive Hemodynamics Workstation, Cardiovascular Engineering Inc.) will be positioned at the carotid and femoral arteries, and CFPWV will be calculated as the mean distance/time between the foot of the carotid and femoral arterial waveforms calculated over >30 heart cycles. Data will be expressed as m/s. Change in CFPWV from baseline to end-intervention will be determined.
Change in Casual (seated, resting) systolic blood pressure | 12 weeks
  Casual (resting, seated) measures of blood pressure (mmHg) will be measured according to American Heart Association/American College of Cardiology guidelines. Briefly, blood pressure will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure. Subjects will be seated quietly with their back supported, feet flat on the floor, and arm at heart level. Casual systolic blood pressure (SBP) will be defined as the average of the three measures. Change in casual SBP from baseline to end-intervention will be determined.

OTHER OUTCOMES:
Change in 24-hour ambulatory blood pressure | 12 weeks
  Brachial artery blood pressure (mmHg) will be measured automatically every 20 minutes for a 24-hour period by an ambulatory blood pressure monitor (Oscar 2, SunTech Medical) validated according to British Hypertension Society Standards. Participants will be outfitted with the ambulatory blood pressure monitor by a trained investigator. The blood pressure cuff will be placed securely on the participant's non-dominant arm. Participants will be given written and verbal instructions on monitor operation. Ambulatory blood pressure recordings will be analyzed for mean 24-hour (averaged over the entire 24-hour period) SBP, and the change in 24-hour SBP from baseline to end-intervention will be determined.
Incidence of enrolled subjects dropping out of the study due to adverse events | 12 weeks
  The rate at which enrolled subjects drop out of the study due to adverse events, as an indicator of the degree to which overt adverse effects can be tolerated by our subjects.
% of prescribed amount of drug that is consumed | 12 weeks
  Adherence to the intervention will be assessed by determining the average % of prescribed study drug that is actually consumed by subjects across the intervention.
Change in serum acetate | 12 weeks
  Venous blood samples will be analyzed for concentrations of acetate using commercially available kit.
Change in gut microbiome composition | 12 weeks
  16S rRNA genes isolated from fecal bacterial DNA (3 fecal swabs) will be amplified at the V4 region and subjected to multiplex Illumina sequencing. Raw sequences will be processed using the Qiita deblur pipeline and assigned taxonomic classification using the feature-classifier/classify-sklearn plugin in QIIME2. Differential abundance across time into the interventions and across groups (acetate vs. placebo) will be analyzed via ANCOM.
Change in Suppression of Brachial Artery Flow-Mediated Dilation by Oxidative Stress | Baseline, 12 weeks
  Suppression of FMDba will be determined as the difference in FMDba (%change units) following 20 minutes of intravenous infusion with vitamin C (0.06 g/kg fat-free mass) vs. following 20 minutes of intravenous infusion with saline. The change in this outcome will be determined from baseline to end-intervention.
Change in Endothelial Cell Markers of Oxidative Stress | 12 weeks
  Endothelial cells will be obtained from an antecubital vein via clinical endovascular biopsy--2 sterile 0.025-inch J-wires will briefly advanced through an intravenous catheter. Cells will be recovered by centrifugation, fixed with formaldehyde, and slides will be prepared and frozen. Slides will be stained for the primary antibody of interest and a complementary fluorescent secondary Alexafluor 647 antibody (Invitrogen). Slides will also be stained for the extracellular domain of vascular endothelial cadherin (Abcam) for positive identification of endothelial phenotype and DAPI for nuclear integrity. Images will be digitally captured and analyzed using Metamorph Software (Universal Imaging Corp). Values will be reported as ratios of subject endothelial cell protein expression to human umbilical vein endothelial cell control cells protein expression. We will determine the change in expression of proteins related to oxidative stress (e.g., nitrotyrosine and NADPH oxidase).

CONTACTS AND LOCATIONS:
Overall Officials: Vienna Brunt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No